CLINICAL TRIAL: NCT06686043
Title: A Phase 2 Study of HPV L1 Vaccine in Combination With Imiquimod and Metformin in Cervical, Vaginal, and Vulvar Cancers
Brief Title: HPV Vaccine, Imiquimod, and Metformin Combination Trial
Acronym: HPV-VIM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Harris Health (Unknown); Dan L Duncan Comprehensive Cancer Center (Unknown); Baylor St. Luke's Medical Center (Other)
Responsible Party: Principal Investigator, Jan Sivert Sunde, DIVISION DIRECTOR, GYNECOLOGIC ONCOLOGY Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-54674
Record Dates: First submitted 2024-11-03; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cervical Carcinoma; Vaginal Carcinoma; Vulvar Carcinoma; HPV (Human Papillomavirus)-Associated Carcinoma
Keywords: metformin; HPV; Imiquimod; Human Papillomavirus 9-valent Vaccine; Recombinant; Cytobrush; cervical cancer; vaginal cancer; vulvar cancer; chemoradiation; tumor; immunotherapy; metastatic; intratumoral; Endometrial cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Papillomavirus Infections; Neoplasms; Neoplasm Metastasis; Endometrial Neoplasms | interventions — Papillomavirus Vaccines; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment group (Experimental): The treatment group will be compared to a historical control. The investigator will evaluate the immune changes within the tumor microenvironment and validate why the combination immunotherapy study elicited such a robust immune response which led to complete resolution of the cancer, in comparison to the standard of care, chemoradiation. In this study, participants will undergo a series of treatment visits during and after radiation therapy to assess the effectiveness of the experimental combination therapy.
  Interventions: Drug: HPV vaccine, Imiquimod, and metformin combination therapy

INTERVENTIONS:
Drug: HPV vaccine, Imiquimod, and metformin combination therapy — Participants in the treatment arm will have visits during the 2nd and 4th weeks of radiation, and then at weeks 8, 10, 12, and 16 after radiation. At each visit, a blood sample will be taken, and tumor cells collected using a cytobrush (or directly from the tumor for vulvar cancer). An HPV vaccine will be injected into the tumor, imiquimod cream will be applied topically, and participants will receive a subcutaneous vaccine shot. They will also take metformin tablets twice daily for two weeks and apply imiquimod cream at home three nights per week. Follow-up PET/CT scans will occur at week 20 and two years post-treatment, with exams every three months for two years.

SUMMARY:
The goal of this clinical trial is to explore whether additional treatments can help strengthen the participant's immune system to fight cancer caused by the Human Papillomavirus (HPV), a virus spread through intimate skin-to-skin contact. The trial will also monitor the safety of these treatments. The main questions it aims to answer are:

Does the combination of treatments help the participant's body fight the cancer more effectively when used alongside standard therapy? What side effects or medical issues arise when using these experimental treatments? Researchers will use three experimental therapies along with the participant's standard treatment to find out if these therapies work better together than standard treatment alone.

Participants will:

Receive HPV vaccinations during the 2nd and 4th week of radiation, and again at weeks 8, 10, 12, and 16 after completing radiation.

Have blood samples taken, tumor cells brushed from the surface, and imiquimod cream applied during each visit.

Take a daily metformin pill and apply an imiquimod suppository three times a week for two weeks after each visit.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine whether stimulating tumor immunity through sequential, targeted intratumoral vaccinations using the FDA-approved quadrivalent HPV-L1 antigen vaccine, in combination with chemotherapy, radiotherapy, pembrolizumab, imiquimod, and metformin, improves outcomes for patients with locally advanced cervical, vaginal, or vulvar carcinoma. The primary objective is to assess the impact of this approach on 24-month progression-free survival when used alongside whole pelvic radiotherapy, chemotherapy, and brachytherapy.

The trial will also monitor the safety and potential side effects of combining intratumoral HPV vaccination with topical imiquimod and oral metformin during and after chemoradiation. Additionally, researchers aim to evaluate specific immune markers to understand how these treatments boost the immune system and enhance the effects of standard care.

Participants will:

Receive intratumoral HPV vaccinations during the 2nd and 4th week of radiation, and after completing radiation at weeks 8, 10, 12, and 16.

Have blood samples taken, tumor cells brushed, and imiquimod cream applied during each visit.

Take a daily metformin pill and apply an imiquimod suppository three times a week for two weeks after each visit.

Throughout the trial, immune biomarker assays will be conducted at the beginning, middle, and end of treatment to measure markers such as CD4, CD8, NK, TNF alpha and beta, IL2, HPV viral load, TGF Beta, Ki67, and IgG. Blood tests will also be done for IgG L1 and L2, E6 and E7, and a CBC, to track immune changes across the three treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed locally advanced or metastatic cervical carcinoma (Stage IB2-IVB), vaginal, or vulvar carcinoma (Stage II-IVB), AND not be considered a primary surgical candidate. Patients offered neoadjuvant therapy may be enrolled if they respond and receive chemoradiation.
* Participants must have measurable disease, per Recist criteria. See Section 12 (Measurement of Effect) for the evaluation of measurable disease. Radiological evaluation shall occur within approximately 30 days prior to enrollment initiation and start of radiation.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Participants must be ≥ 18 years of age
* Participants must have adequate organ function within 28 days of registration, defined as follows: - Absolute neutrophil count ≥ 1,500/µL - Platelets ≥ 100,000/µL - Hemoglobin ≥ 9 g/dL - Serum creatinine ≤ 1.5 x upper limit of normal (ULN) - Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN - Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Participants receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy.
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Female participants of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. Females of non-childbearing potential is defined as follows (by other than medical reasons): - ≥45 years of age and has not had menses for >1 year, post-hysterectomy, post-bilateral oophorectomy, post external beam radiation of 6 Gy to the pelvis, or post-tubal ligation.
* Participants must agree to not breastfeed during the study.
* Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent
* Participants must be eligible for chemoradiation treatment in the opinion of the treating investigator.
* Participants who are HIV+ must have CD4 counts >200/dL and demonstrate documented Highly active antiretroviral therapy (HAART) compliance m. Participant must have CT (chest/abdomen/pelvis) or PET-CT, within 56 days of registration.
* Participants must be newly diagnosed.
* Standard chemoradiation using external beam radiation therapy (EBRT) and brachytherapy is permitted for cervical or vaginal carcinoma, and chemoradiation with EBRT for vulvar carcinoma. A lesion must be readily accessible for intratumoral tumor injection.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Patients who have untreated, new or progressive brain metastases or leptomeningeal disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because cervical carcinoma or vulva carcinoma patients have undergone treatment rendering the patient infertile. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cervical carcinoma or vulva carcinoma, breastfeeding should be discontinued.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-08-23 (Estimated); Study Completion 2028-08-23 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  Progression-free survival at 24 months will be collected for all patients.

SECONDARY OUTCOMES:
Common Toxicity Criteria (CTC) | 24 months
  Discontinuation rate of medications during treatments due to potential side effects
Identify Immune changes | 24 months
  Immune biomarker assays will be taken at the beginning, middle, and end of the treatment to measure the following markers: CD4, CD8, NK, TNF alpha and beta, IL2, HPV viral load, TGF Beta, Ki67, IGg. We will also do blood tests to test for IGg L1 and L2, E6 and E7 and a CBC. These markers combined were chosen to identify specific immune changes of the three medication treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan S Sunde, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor St. Luke's Medical Center- Dan L. Duncan Comprehensive Cancer Center, Houston, Texas
  - Harris Health Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The study team will deposit deidentified data in on-line database
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of study completion.
Access Criteria: Public access database
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Tantipalakorn C, Robertson G, Marsden DE, Gebski V, Hacker NF. Outcome and patterns of recurrence for International Federation of Gynecology and Obstetrics (FIGO) stages I and II squamous cell vulvar cancer. Obstet Gynecol. 2009 Apr;113(4):895-901. doi: 10.1097/AOG.0b013e31819b413f. PMID 19305336
- [Background] Reedy M, Jonnalagadda S, Palle K. Case Report: Intra-Tumoral Vaccinations of Quadrivalent HPV-L1 Peptide Vaccine With Topical TLR-7 Agonist Following Recurrence: Complete Resolution of HPV-HR-Associated Gynecologic Squamous Cell Carcinomas in Two Patients. Pathol Oncol Res. 2021 Dec 20;27:1609922. doi: 10.3389/pore.2021.1609922. eCollection 2021. PMID 34987310
- [Background] Mondini M, Nizard M, Tran T, Mauge L, Loi M, Clemenson C, Dugue D, Maroun P, Louvet E, Adam J, Badoual C, Helley D, Dransart E, Johannes L, Vozenin MC, Perfettini JL, Tartour E, Deutsch E. Synergy of Radiotherapy and a Cancer Vaccine for the Treatment of HPV-Associated Head and Neck Cancer. Mol Cancer Ther. 2015 Jun;14(6):1336-45. doi: 10.1158/1535-7163.MCT-14-1015. Epub 2015 Apr 1. PMID 25833837
- [Background] Mu J, Lei L, Zheng Y, Li D, Li J, Fu Y, Wang G, Liu Y. Comparative study of subcutaneous, intramuscular, and oral administration of bovine pathogenic Escherichia coli bacterial ghost vaccine in mice. Front Immunol. 2022 Nov 14;13:1008131. doi: 10.3389/fimmu.2022.1008131. eCollection 2022. PMID 36451816
- [Background] Afzal MZ, Mercado RR, Shirai K. Efficacy of metformin in combination with immune checkpoint inhibitors (anti-PD-1/anti-CTLA-4) in metastatic malignant melanoma. J Immunother Cancer. 2018 Jul 2;6(1):64. doi: 10.1186/s40425-018-0375-1. PMID 29966520
- [Background] Wu Z, Zhang C, Najafi M. Targeting of the tumor immune microenvironment by metformin. J Cell Commun Signal. 2022 Sep;16(3):333-348. doi: 10.1007/s12079-021-00648-w. Epub 2021 Oct 5. PMID 34611852
- [Background] Ma R, Yi B, Riker AI, Xi Y. Metformin and cancer immunity. Acta Pharmacol Sin. 2020 Nov;41(11):1403-1409. doi: 10.1038/s41401-020-00508-0. Epub 2020 Aug 31. PMID 32868904
- [Background] Tselikas L, Dardenne A, de Baere T, Faron M, Ammari S, Farhane S, Suzzoni S, Danlos FX, Raoult T, Susini S, Al Shatti N, Mouraud S, Deschamps F, Kobe A, Delpla A, Roux C, Baldini C, Soria JC, Barlesi F, Massard C, Robert C, Champiat S, Marabelle A. Feasibility, safety and efficacy of human intra-tumoral immuno-therapy. Gustave Roussy's initial experience with its first 100 patients. Eur J Cancer. 2022 Sep;172:1-12. doi: 10.1016/j.ejca.2022.05.024. Epub 2022 Jun 18. PMID 35724442
- [Background] van de Sande AJM, Kengsakul M, Koeneman MM, Jozwiak M, Gerestein CG, Kruse AJ, van Esch EMG, de Vos van Steenwijk PJ, Muntinga CLP, Bramer WM, van Doorn HC, van Kemenade FJ, van Beekhuizen HJ. The efficacy of topical imiquimod in high-grade cervical intraepithelial neoplasia: A systematic review and meta-analysis. Int J Gynaecol Obstet. 2024 Jan;164(1):66-74. doi: 10.1002/ijgo.14953. Epub 2023 Jun 23. PMID 37350560
- [Background] Rosales R, Lopez-Contreras M, Rosales C, Magallanes-Molina JR, Gonzalez-Vergara R, Arroyo-Cazarez JM, Ricardez-Arenas A, Del Follo-Valencia A, Padilla-Arriaga S, Guerrero MV, Pirez MA, Arellano-Fiore C, Villarreal F. Regression of human papillomavirus intraepithelial lesions is induced by MVA E2 therapeutic vaccine. Hum Gene Ther. 2014 Dec;25(12):1035-49. doi: 10.1089/hum.2014.024. PMID 25275724
- [Background] Marei A, Nofal A, Alakad R, Abdel-Hady A. Combined bivalent human papillomavirus vaccine and Candida antigen versus Candida antigen alone in the treatment of recalcitrant warts. J Cosmet Dermatol. 2020 Mar;19(3):758-762. doi: 10.1111/jocd.13077. Epub 2019 Jul 22. PMID 31328869
- [Background] Mori V, DuComb EA, Wagner S, Khan F, Bates JHT, Kinsey CM. Visualizing intratumoral injections in lung tumors by endobronchial ultrasound. J Cancer. 2023 Feb 22;14(4):544-553. doi: 10.7150/jca.81793. eCollection 2023. PMID 37057292
- [Background] Kidner TB, Morton DL, Lee DJ, Hoban M, Foshag LJ, Turner RR, Faries MB. Combined intralesional Bacille Calmette-Guerin (BCG) and topical imiquimod for in-transit melanoma. J Immunother. 2012 Nov-Dec;35(9):716-20. doi: 10.1097/CJI.0b013e31827457bd. PMID 23090081
- [Background] Omland SH, Ejlertsen JS, Krustrup D, Christensen RL, Svane IM, Olesen UH, Haedersdal M. Feasibility of Intratumoral Anti-PD1 as Treatment of Human Basal Cell Carcinoma: An Explorative Study with Adjuvant Ablative Fractional Laser. Cancers (Basel). 2022 Nov 25;14(23):5815. doi: 10.3390/cancers14235815. PMID 36497301
- [Background] Ponce S, Cedres S, Ricordel C, Isambert N, Viteri S, Herrera-Juarez M, Martinez-Marti A, Navarro A, Lederlin M, Serres X, Zugazagoitia J, Vetrhus S, Jaderberg M, Hansen TB, Levitsky V, Paz-Ares L. ONCOS-102 plus pemetrexed and platinum chemotherapy in malignant pleural mesothelioma: a randomized phase 2 study investigating clinical outcomes and the tumor microenvironment. J Immunother Cancer. 2023 Sep;11(9):e007552. doi: 10.1136/jitc-2023-007552. PMID 37661097
- [Background] Luke JJ, Piha-Paul SA, Medina T, Verschraegen CF, Varterasian M, Brennan AM, Riese RJ, Sokolovska A, Strauss J, Hava DL, Janku F. Phase I Study of SYNB1891, an Engineered E. coli Nissle Strain Expressing STING Agonist, with and without Atezolizumab in Advanced Malignancies. Clin Cancer Res. 2023 Jul 5;29(13):2435-2444. doi: 10.1158/1078-0432.CCR-23-0118. PMID 37227176
- [Background] Meric-Bernstam F, Sweis RF, Kasper S, Hamid O, Bhatia S, Dummer R, Stradella A, Long GV, Spreafico A, Shimizu T, Steeghs N, Luke JJ, McWhirter SM, Muller T, Nair N, Lewis N, Chen X, Bean A, Kattenhorn L, Pelletier M, Sandhu S. Combination of the STING Agonist MIW815 (ADU-S100) and PD-1 Inhibitor Spartalizumab in Advanced/Metastatic Solid Tumors or Lymphomas: An Open-Label, Multicenter, Phase Ib Study. Clin Cancer Res. 2023 Jan 4;29(1):110-121. doi: 10.1158/1078-0432.CCR-22-2235. PMID 36282874
- [Background] Babiker H, Borazanci E, Subbiah V, Agarwala S, Algazi A, Schachter J, Lotem M, Maurice-Dror C, Hendler D, Rahimian S, Minderman H, Haymaker C, Mahadevan D, Bernatchez C, Murthy R, Hultsch R, Kaplan N, Woodhead G, Hennemeyer C, Chunduru S, Anderson PM, Diab A, Puzanov I. Tilsotolimod Exploits the TLR9 Pathway to Promote Antigen Presentation and Type 1 IFN Signaling in Solid Tumors: A Multicenter International Phase I/II Trial (ILLUMINATE-101). Clin Cancer Res. 2022 Dec 1;28(23):5079-5087. doi: 10.1158/1078-0432.CCR-21-4486. PMID 35917516
- [Background] Bonvalot S, Rutkowski PL, Thariat J, Carrere S, Ducassou A, Sunyach MP, Agoston P, Hong A, Mervoyer A, Rastrelli M, Moreno V, Li RK, Tiangco B, Herraez AC, Gronchi A, Mangel L, Sy-Ortin T, Hohenberger P, de Baere T, Le Cesne A, Helfre S, Saada-Bouzid E, Borkowska A, Anghel R, Co A, Gebhart M, Kantor G, Montero A, Loong HH, Verges R, Lapeire L, Dema S, Kacso G, Austen L, Moureau-Zabotto L, Servois V, Wardelmann E, Terrier P, Lazar AJ, Bovee JVMG, Le Pechoux C, Papai Z. NBTXR3, a first-in-class radioenhancer hafnium oxide nanoparticle, plus radiotherapy versus radiotherapy alone in patients with locally advanced soft-tissue sarcoma (Act.In.Sarc): a multicentre, phase 2-3, randomised, controlled trial. Lancet Oncol. 2019 Aug;20(8):1148-1159. doi: 10.1016/S1470-2045(19)30326-2. Epub 2019 Jul 8. PMID 31296491
- [Background] Spalato-Ceruso M, Bouteiller F, Guegan JP, Toulmonde M, Bessede A, Kind M, Cousin S, Buy X, Palussiere J, Le Loarer F, Dadone-Montaudie B, Pulido M, Italiano A. Pembrolizumab combined with low-dose cyclophosphamide and intra-tumoral injection of the toll-like receptor 4 agonist G100 in patients with advanced pretreated soft tissue sarcoma: results from the PEMBROSARC basket study. J Hematol Oncol. 2022 Oct 27;15(1):157. doi: 10.1186/s13045-022-01377-2. PMID 36303228
- [Background] Chawla SP, Tellez WA, Chomoyan H, Valencia C, Ahari A, Omelchenko N, Makrievski S, Brigham DA, Chua-Alcala V, Quon D, Moradkhani A, Gordon EM. Activity of TNT: a phase 2 study using talimogene laherparepvec, nivolumab and trabectedin for previously treated patients with advanced sarcomas (NCT# 03886311). Front Oncol. 2023 May 10;13:1116937. doi: 10.3389/fonc.2023.1116937. eCollection 2023. PMID 37234994
- [Background] Miller M, Kim NH, Thosani MK, Moser JC. Use of Talimogene Laherparepvec to Treat Cutaneous Squamous Cell Carcinoma in a Renal Transplant Patient. Case Rep Dermatol. 2023 Jun 13;15(1):99-104. doi: 10.1159/000530851. eCollection 2023 Jan-Dec. PMID 37383323
- [Background] Nguyen VP, Campbell KM, Nowicki TS, Elumalai N, Medina E, Baselga-Carretero I, DiNome ML, Chang HR, Oseguera DK, Ribas A, Glaspy JA. A Pilot Study of Neoadjuvant Nivolumab, Ipilimumab, and Intralesional Oncolytic Virotherapy for HER2-negative Breast Cancer. Cancer Res Commun. 2023 Aug 23;3(8):1628-1637. doi: 10.1158/2767-9764.CRC-23-0145. eCollection 2023 Aug. PMID 37621406
- [Background] Soliman H, Hogue D, Han H, Mooney B, Costa R, Lee MC, Niell B, Williams A, Chau A, Falcon S, Soyano A, Armaghani A, Khakpour N, Weinfurtner RJ, Hoover S, Kiluk J, Laronga C, Rosa M, Khong H, Czerniecki B. Oncolytic T-VEC virotherapy plus neoadjuvant chemotherapy in nonmetastatic triple-negative breast cancer: a phase 2 trial. Nat Med. 2023 Feb;29(2):450-457. doi: 10.1038/s41591-023-02210-0. Epub 2023 Feb 9. PMID 36759673
- [Background] Margalit O, Lieberman S, Redinsky I, Halparin S, Honig N, Raskin S, Ben-Ayun M, Shacham-Shmueli E, Halpern N, Urban D, Ackerstein A, Shulman K, Ben-Ami E, Semenisty V, Purim O, Yarom N, Golan T, Boursi B, Appel S, Symon Z, Berger R, Mauro D, Krieg AM, Lawrence YR. Combination Treatment of Intratumoral Vidutolimod, Radiosurgery, Nivolumab, and Ipilimumab for Microsatellite Stable Colorectal Carcinoma With Liver Metastases. Clin Colorectal Cancer. 2023 Dec;22(4):442-449.e1. doi: 10.1016/j.clcc.2023.08.004. Epub 2023 Aug 9. PMID 37657954
- [Background] Heo J, Liang JD, Kim CW, Woo HY, Shih IL, Su TH, Lin ZZ, Yoo SY, Chang S, Urata Y, Chen PJ. Safety and dose escalation of the targeted oncolytic adenovirus OBP-301 for refractory advanced liver cancer: Phase I clinical trial. Mol Ther. 2023 Jul 5;31(7):2077-2088. doi: 10.1016/j.ymthe.2023.04.006. Epub 2023 Apr 14. PMID 37060176
- [Background] Gogenur M, Balsevicius L, Bulut M, Colak N, Justesen TF, Fiehn AK, Jensen MB, Host-Rasmussen K, Cappelen B, Gaggar S, Tajik A, Zahid JA, Bennedsen ALB, D'Ondes TDB, Raskov H, Saekmose SG, Hansen LB, Salanti A, Brix S, Gogenur I. Neoadjuvant intratumoral influenza vaccine treatment in patients with proficient mismatch repair colorectal cancer leads to increased tumor infiltration of CD8+ T cells and upregulation of PD-L1: a phase 1/2 clinical trial. J Immunother Cancer. 2023 May;11(5):e006774. doi: 10.1136/jitc-2023-006774. PMID 37172969
- [Background] Curti BD, Richards J, Hyngstrom JR, Daniels GA, Faries M, Feun L, Margolin KA, Hallmeyer S, Grose M, Zhang Y, Li A, Andtbacka RHI. Intratumoral oncolytic virus V937 plus ipilimumab in patients with advanced melanoma: the phase 1b MITCI study. J Immunother Cancer. 2022 Dec;10(12):e005224. doi: 10.1136/jitc-2022-005224. PMID 36564126
- [Background] Shimbo T, Yoshida K, Nakata M, Kobata K, Ogawa T, Kihara A, Sato C, Hori A, Takeno S, Yoshioka H, Akiyama H, Nihei K. KORTUC, a novel hydrogen peroxide-based radiosensitizer for the enhancement of brachytherapy in patients with unresectable recurrent uterine cervical cancer. Oncol Lett. 2023 Jul 20;26(3):378. doi: 10.3892/ol.2023.13964. eCollection 2023 Sep. PMID 37559582
- [Background] Yoshikawa R, Inoue J, Iwasaki R, Terauchi M, Fujii Y, Ohta M, Hasegawa T, Mizuno R, Mori T, Inazawa J. Therapeutic applications of local injection of hsa-miR-634 into canine spontaneous malignant melanoma tumors. Cancer Gene Ther. 2023 Nov;30(11):1524-1529. doi: 10.1038/s41417-023-00656-5. Epub 2023 Aug 8. PMID 37553484
- [Background] Nobuoka D, Yoshikawa T, Takahashi M, Iwama T, Horie K, Shimomura M, Suzuki S, Sakemura N, Nakatsugawa M, Sadamori H, Yagi T, Fujiwara T, Nakatsura T. Intratumoral peptide injection enhances tumor cell antigenicity recognized by cytotoxic T lymphocytes: a potential option for improvement in antigen-specific cancer immunotherapy. Cancer Immunol Immunother. 2013 Apr;62(4):639-52. doi: 10.1007/s00262-012-1366-6. Epub 2012 Nov 11. PMID 23143746
- [Background] Ishida E, Lee J, Campbell JS, Chakravarty PD, Katori Y, Ogawa T, Johnson L, Mukhopadhyay A, Faquin WC, Lin DT, Wirth LJ, Pierce RH, Pai SI. Intratumoral delivery of an HPV vaccine elicits a broad anti-tumor immune response that translates into a potent anti-tumor effect in a preclinical murine HPV model. Cancer Immunol Immunother. 2019 Aug;68(8):1273-1286. doi: 10.1007/s00262-019-02357-1. Epub 2019 Jun 26. PMID 31243491
- [Background] Gustafson LW, Gade M, Blaakaer J. Vulval cancer and HPV vaccination in recurrent disease. Clin Case Rep. 2014 Dec;2(6):243-6. doi: 10.1002/ccr3.93. Epub 2014 Nov 17. PMID 25548622
- [Background] Garland SM, Paavonen J, Jaisamrarn U, Naud P, Salmeron J, Chow SN, Apter D, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Limson G, Schwarz TF, Poppe WA, Bosch FX, de Carvalho NS, Germar MJ, Peters K, Del Rosario-Raymundo MR, Catteau G, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Prior human papillomavirus-16/18 AS04-adjuvanted vaccination prevents recurrent high grade cervical intraepithelial neoplasia after definitive surgical therapy: Post-hoc analysis from a randomized controlled trial. Int J Cancer. 2016 Dec 15;139(12):2812-2826. doi: 10.1002/ijc.30391. Epub 2016 Sep 9. PMID 27541373
- [Background] Zhang X, Wang Y, Lv X, Wang F, Zhou Q, Zhang F, Zhang M, Chen J. Intratumoral injection of oncolytic virus (H101) in combination with concurrent chemoradiotherapy for locally advanced cervical cancer. Int J Gynecol Cancer. 2023 Jul 3;33(7):1051-1056. doi: 10.1136/ijgc-2022-003914. PMID 37208018
- [Background] Morris ZS, Guy EI, Francis DM, Gressett MM, Werner LR, Carmichael LL, Yang RK, Armstrong EA, Huang S, Navid F, Gillies SD, Korman A, Hank JA, Rakhmilevich AL, Harari PM, Sondel PM. In Situ Tumor Vaccination by Combining Local Radiation and Tumor-Specific Antibody or Immunocytokine Treatments. Cancer Res. 2016 Jul 1;76(13):3929-41. doi: 10.1158/0008-5472.CAN-15-2644. Epub 2016 May 6. PMID 27197149
- [Background] Huang L, Ge X, Liu Y, Li H, Zhang Z. The Role of Toll-like Receptor Agonists and Their Nanomedicines for Tumor Immunotherapy. Pharmaceutics. 2022 Jun 10;14(6):1228. doi: 10.3390/pharmaceutics14061228. PMID 35745800
- [Background] Trutnovsky G, Reich O, Joura EA, Holter M, Ciresa-Konig A, Widschwendter A, Schauer C, Bogner G, Jan Z, Boandl A, Kalteis MS, Regauer S, Tamussino K. Topical imiquimod versus surgery for vulvar intraepithelial neoplasia: a multicentre, randomised, phase 3, non-inferiority trial. Lancet. 2022 May 7;399(10337):1790-1798. doi: 10.1016/S0140-6736(22)00469-X. Epub 2022 Apr 25. PMID 35483400
- [Background] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Background] Terlou A, van Seters M, Ewing PC, Aaronson NK, Gundy CM, Heijmans-Antonissen C, Quint WG, Blok LJ, van Beurden M, Helmerhorst TJ. Treatment of vulvar intraepithelial neoplasia with topical imiquimod: seven years median follow-up of a randomized clinical trial. Gynecol Oncol. 2011 Apr;121(1):157-62. doi: 10.1016/j.ygyno.2010.12.340. Epub 2011 Jan 15. PMID 21239049
- [Background] Tran CA, Lynch KT, Meneveau MO, Katyal P, Olson WC, Slingluff CL Jr. Intratumoral IFN-gamma or topical TLR7 agonist promotes infiltration of melanoma metastases by T lymphocytes expanded in the blood after cancer vaccine. J Immunother Cancer. 2023 Feb;11(2):e005952. doi: 10.1136/jitc-2022-005952. PMID 36746511
- [Background] Scholch S, Rauber C, Weitz J, Koch M, Huber PE. TLR activation and ionizing radiation induce strong immune responses against multiple tumor entities. Oncoimmunology. 2015 May 7;4(11):e1042201. doi: 10.1080/2162402X.2015.1042201. eCollection 2015 Nov. PMID 26451314
- [Background] Zhai D, An D, Wan C, Yang K. Radiotherapy: Brightness and darkness in the era of immunotherapy. Transl Oncol. 2022 May;19:101366. doi: 10.1016/j.tranon.2022.101366. Epub 2022 Feb 23. PMID 35219093
- [Background] Cho JH, Lee HJ, Ko HJ, Yoon BI, Choe J, Kim KC, Hahn TW, Han JA, Choi SS, Jung YM, Lee KH, Lee YS, Jung YJ. The TLR7 agonist imiquimod induces anti-cancer effects via autophagic cell death and enhances anti-tumoral and systemic immunity during radiotherapy for melanoma. Oncotarget. 2017 Apr 11;8(15):24932-24948. doi: 10.18632/oncotarget.15326. PMID 28212561
- [Background] Cadena A, Cushman TR, Anderson C, Barsoumian HB, Welsh JW, Cortez MA. Radiation and Anti-Cancer Vaccines: A Winning Combination. Vaccines (Basel). 2018 Jan 30;6(1):9. doi: 10.3390/vaccines6010009. PMID 29385680
- [Background] Chuang CM, Monie A, Hung CF, Wu TC. Treatment with imiquimod enhances antitumor immunity induced by therapeutic HPV DNA vaccination. J Biomed Sci. 2010 Apr 28;17(1):32. doi: 10.1186/1423-0127-17-32. PMID 20426849
- [Background] Bellone S, El-Sahwi K, Cocco E, Casagrande F, Cargnelutti M, Palmieri M, Bignotti E, Romani C, Silasi DA, Azodi M, Schwartz PE, Rutherford TJ, Pecorelli S, Santin AD. Human papillomavirus type 16 (HPV-16) virus-like particle L1-specific CD8+ cytotoxic T lymphocytes (CTLs) are equally effective as E7-specific CD8+ CTLs in killing autologous HPV-16-positive tumor cells in cervical cancer patients: implications for L1 dendritic cell-based therapeutic vaccines. J Virol. 2009 Jul;83(13):6779-89. doi: 10.1128/JVI.02443-08. Epub 2009 Apr 22. PMID 19386711
- [Background] Marabelle A, Kohrt H, Caux C, Levy R. Intratumoral immunization: a new paradigm for cancer therapy. Clin Cancer Res. 2014 Apr 1;20(7):1747-56. doi: 10.1158/1078-0432.CCR-13-2116. PMID 24691639
- [Background] Wiemann B, Starnes CO. Coley's toxins, tumor necrosis factor and cancer research: a historical perspective. Pharmacol Ther. 1994;64(3):529-64. doi: 10.1016/0163-7258(94)90023-x. PMID 7724661
- [Background] Gjyshi O, Grippin A, Andring L, Jhingran A, Lin LL, Bronk J, Eifel PJ, Joyner MM, Sastry JK, Yoshida-Court K, Solley TN, Napravnik TC, O'Hara MP, Hegde VL, Colbert LE, Klopp AH. Circulating neutrophils and tumor-associated myeloid cells function as a powerful biomarker for response to chemoradiation in locally advanced cervical cancer. Clin Transl Radiat Oncol. 2023 Jan 11;39:100578. doi: 10.1016/j.ctro.2023.100578. eCollection 2023 Mar. PMID 36935860
- [Background] Dorta-Estremera S, Colbert LE, Nookala SS, Yanamandra AV, Yang G, Delgado A, Mikkelson M, Eifel P, Jhingran A, Lilie LL, Welsh J, Schmeler K, Sastry JK, Klopp A. Kinetics of Intratumoral Immune Cell Activation During Chemoradiation for Cervical Cancer. Int J Radiat Oncol Biol Phys. 2018 Nov 1;102(3):593-600. doi: 10.1016/j.ijrobp.2018.06.404. Epub 2018 Jul 12. PMID 30017792
- [Background] Dorta-Estremera S, Nehete PN, Yang G, He H, Nehete BP, Shelton KA, Barry MA, Sastry KJ. Minimally invasive monitoring of CD4 T cells at multiple mucosal tissues after intranasal vaccination in rhesus macaques. PLoS One. 2017 Dec 8;12(12):e0188807. doi: 10.1371/journal.pone.0188807. eCollection 2017. PMID 29220358
- [Background] McKinnon LR, Hughes SM, De Rosa SC, Martinson JA, Plants J, Brady KE, Gumbi PP, Adams DJ, Vojtech L, Galloway CG, Fialkow M, Lentz G, Gao D, Shu Z, Nyanga B, Izulla P, Kimani J, Kimwaki S, Bere A, Moodie Z, Landay AL, Passmore JA, Kaul R, Novak RM, McElrath MJ, Hladik F. Optimizing viable leukocyte sampling from the female genital tract for clinical trials: an international multi-site study. PLoS One. 2014 Jan 15;9(1):e85675. doi: 10.1371/journal.pone.0085675. eCollection 2014. PMID 24454917
- [Background] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- [Background] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124

DOCUMENTS (1):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT06686043/Prot_000.pdf